CLINICAL TRIAL: NCT06578195
Title: ASSESS ALL ALS - Longitudinal Biomarker Study for Symptomatic ALS and Control Participants
Brief Title: ASSESS ALL ALS Study
Status: Recruiting | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Foundation for the National Institutes of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2024P001132; 1OT2NS136938 (NIH); 1OT2NS136939 (NIH)
Record Dates: First submitted 2024-08-20; First posted 2024-08-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; biomarker; observational
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic ALS on-site participants: Symptomatic ALS Participants who are completing on-site visits at one of the 35 participating ALL ALS sites.
- Symptomatic ALS off-site (remote) participants: Symptomatic ALS Participants who are completing visits study visits remotely through video-conferencing. Home Phlebotomy is being used to collect blood from these participants.
- Control participants: Control participants who do not have a diagnosis of ALS , Progressive Muscular Atrophy (PMA) or Primary Lateral Sclerosis (PLS). These participants complete on-site visits.

SUMMARY:
The ALL ALS Clinical Research Consortium is establishing research to collect a wide range of samples, clinical information and measurements from Amyotrophic Lateral Sclerosis (ALS) symptomatic, ALS gene carriers and control cohorts. This consortium is being funded by the National Institutes of Health/National Institute of Neurological Disorders and Stroke (NIH/NINDS) and managed by two clinical coordinating centers (CCC) at Barrow Neurological Institute and Massachusetts General Hospital. The clinical sites are distributed across the country, and led by a group of collaborative principal investigators. Once data and samples are collected and harmonized, it will be made available to research community for future research into ALS and related neurological diseases.

ASSESS protocol is specific for symptomatic ALS and control participants. This protocol includes both on-site and off-site(remote) participants. The participants will be followed for 24 months (2 years), and will include collection of medical history, clinical outcomes, and blood samples once in 4 months. Additionally, the participants will complete patient reported outcomes and speech recordings once a month. Participants who are coming into clinic may also provide optional Cerebrospinal Fluid (CSF) samples.

ELIGIBILITY:
Inclusion Criteria for ALS participants:

1. Age 18 years or older
2. Capable of providing informed consent
3. Willing to follow study procedures
4. Diagnosis of ALS by a physician
5. Access to a smartphone, computer or tablet, and internet (need not be in the home - access to a public library or other available computer with internet connection is sufficient)

Inclusion Criteria for control participants:

1. Age 18 years or older
2. Capable of providing informed consent
3. Willing to follow study procedures
4. No diagnosis of ALS , Progressive Muscular Atrophy (PMA) or Primary Lateral Sclerosis (PLS)
5. No history of familial ALS/Frontotemporal Dementia (FTD) in a close family member** unless the participant has previously tested negative for the known causative ALS genes. Participants with a family history of singleton ALS are permitted to enroll.

   * ** Defined by the presence of a known ALS causative gene such as C9orf72 in a family member or a family history suggestive of an inherited ALS/FTD syndrome defined by two family members with a history of ALS and/or FTD.
6. Access to a smartphone, computer or tablet, and internet (need not be in the home - access to a public library or other available computer with internet connection is sufficient)

Exclusion Criteria for all participants:

1. Significant cognitive impairment, clinical dementia, or unstable psychiatric illness, including psychosis, active suicidal ideation, suicide attempt, or untreated major depression <= 90 days of screening, that would interfere with the study procedure, according to Investigator's judgement.
2. Clinically significant unstable medical condition (other than ALS) (e.g., cardiovascular instability, systemic infection, untreated thyroid dysfunction, malignant and potentially progressive cancer) that would render the participant unlikely to be able to complete 12 months of follow-up, according to Investigator's judgment.

Exclusion Criteria for participants undergoing optional Lumbar Puncture

1. Medically unable to undergo lumbar puncture (LP) as determined by the site investigator (i.e., bleeding disorder, a skin infection at or near the LP site, known or suspected intracranial or intraspinal tumor or other cause of increased intracranial pressure).
2. Allergy to Lidocaine or other local anesthetic agents.
3. Use of anticoagulant medication or antiplatelet medications (aside from aspirin 81 mg) that cannot be safely withheld prior to lumbar puncture.
4. Blood dyscrasia, abnormal bleeding diathesis, or the use of dialysis for renal failure.
5. Current pregnancy based on participant self-report
6. Clinical judgement of the site investigator that the participant would be unable to undergo multiple lumbar punctures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An initial cohort of approximately 2000 to 3000 participants will be recruited for this study. This includes at least 1600 symptomatic ALS participants (Cohort 1) and at least 450 control participants (Cohort 2). Though the exact percentages of in-clinic and remote participants are unknown at this time, it is anticipated that approximately 600 of the symptomatic ALS participants and 450 of the control participants will be recruited from the site clinic or local ALS community and will be coming to the sites for study visits. These numbers may differ substantially from the final enrollment numbers based on preference of participants enrolling in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-07-25 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) | Baseline, 4, 8, 12, 16, 20 and 24 months for ALS participants only.
  Questionnaire administered by a clinician that includes a series of questions about participants' ability to function in certain daily activities. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
ALS Functional Rating Scale-Revised Self entry (ALSFRS-RSE) | Baseline, 2, 4 ,6, 8, 10, 12, 14,16, 18,20, 22 and 24 months for ALS participants only
  Questionnaires completed by participants that includes questions about participants ability to function in certain daily activities. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.

SECONDARY OUTCOMES:
ALS Impairment Multidomain scale (AIMS) | 1, 3, 5,7,9,11,13,15,17,19,21 and 23 months from baseline for ALS participants only
  Questionnaires completed by participants that assess severity of the ALS disease
Social Determinants of Health | Months 3 and 4 for all cohorts
  Questionnaires completed by participants that includes questions about non-medical factors that affect health outcomes
Environmental History | Month 1 for all cohorts
  Questionnaires completed by participants that includes questions about environmental exposures such as chemicals, smoking, alcohol etc.
Cognitive assessment (ECAS) | Baseline, 12 and 24 months for all cohorts
  ECAS is a multi-domain assessment administered by study staff, to evaluate different aspects of cognitive function
Vital Capacity | Baseline, 4,8,12,16,20 and 24 months for on-site ALS participants; Baseline, 12 and 24 months for control participants
  Change in respiratory function over time as measured by Slow Vital Capacity (SVC).
Digital Speech Assessment | Baseline, and monthly (at month 1,2, 3 through month 24 from baseline)
  Participants will be asked to record voice samples at home once a month using a digital application installed on their device.
HHD of 3 hand muscles bilaterally | Baseline, 4,8,12,16,20 and 24 months for on-site ALS participants; Baseline, 12 and 24 months for control participants
  Hand-held dynamometry (HHD) will be used as a quantitative measure of muscle strength for the three intrinsic hand muscles, bilaterally

CONTACTS AND LOCATIONS:
Locations (32):
- United States (31):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - University of California San Diego, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Hospital For Special Care, New Britain, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Nih/Ninds, Bethseda, Maryland
  - Massachusetts General Brigham, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Colombus, Ohio
  - Providence ALS Center, Portland, Oregon
  - Penn State Health, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Texas Neurology, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- CHALS-CCT, University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico, Puerto Rico